CLINICAL TRIAL: NCT05534061
Title: Motivational Enhancement to Augment Contingency Management for SARS-CoV-2 Testing and Vaccination Utilization Among Syringe Exchange Clients
Brief Title: Motivation, Syringe Exchange, and COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 11162020.013b; 1U01DA055982-01 (NIH)
Record Dates: First submitted 2022-09-07; First posted 2022-09-09 (Actual); Results first posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-01

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Connect2Test Intervention + Contingency Management (Experimental): $10 financial incentive for vaccination and $10 financial incentive for testing plus a brief feedback-based motivational enhancement intervention.
  Interventions: Behavioral: Connect2Test
- Contingency Management Alone (Active Comparator): $10 financial incentive for vaccination and $10 financial incentive for testing.
  Interventions: Behavioral: Connect2Test

INTERVENTIONS:
Behavioral: Connect2Test — Brief motivational enhancement intervention to improve the likelihood of testing and vaccination among syringe exchange clients
  Other Names: Motivational Enhancement

SUMMARY:
People who inject drugs (PWIDs) are highly vulnerable to SARS-CoV-2 infection and to the disease caused by SARS-CoV-2, coronavirus disease 2019 (COVID-19), however, rates of SARS-CoV-2 testing and vaccination uptake -vital to mitigating the spread of COVID-19 and achieving herd immunity - are lower among PWIDs compared to the general population. Building on our Phase I Rapid Acceleration of Diagnostics project, which found that contingency management (CM) increased testing utilization among PWIDs, the proposed project evaluates the comparative effectiveness of CM versus CM plus a brief motivational enhancement intervention on SARS-CoV-2 testing and vaccination uptake among PWIDs. This project has the potential to reduce COVID-19 health disparities among PWIDs and to decrease population level COVID-19 morbidity and mortality.

DETAILED DESCRIPTION:
This study uses contingency management, specifically $10 financial incentives for participation in SARS-CoV-2 testing and $10 for participating in COVID-19 vaccination. It also uses a motivational enhancement intervention which is a brief conversation with clients to improve intrinsic motivation for testing and vaccination. Thus, the clinical trials portion of this study is a randomized control trial (N = 349) in which 177 participants will be assigned to contingency management plus the Connect2Test intervention and 172 will be assigned to the contingency management alone (i.e. services as usual). There will be a per site quota to ensure there are relatively equivalent numbers of participants per site to avoid site-specific biases. The data collection software (e.g., Qualtrics, PowerBI) will randomly assign individuals to condition in real time, after a participant consents to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 and older, understand English

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 349 (Actual)
Dates: Start 2022-08-08 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
In line with funding requirements, we will share data with our data coordination center and the national institutes of health
Supporting Information: Study Protocol, SAP, ICF
URL: https://radx-up.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Connect2Test Intervention + Contingency Management | Contingency Management Alone
Started | 177 | 172
Completed | 177 | 172
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Connect2Test Intervention + Contingency Management | Contingency Management Alone | Total
Number analyzed (Participants) | 177 | 172 | 349
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.60 (11.23) | 45.19 (10.80) | 43.92 (11.11)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 53 | 51 | 104
  Male | 89 | 88 | 177
  Non-binary | 2 | 4 | 6
  Bigender | 0 | 2 | 2
  None of the listed categories | 2 | 2 | 4
  Unknown or not reported | 31 | 25 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 8 | 14
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 4 | 1 | 5
  Black or African American | 0 | 4 | 4
  White | 109 | 113 | 222
  More than one race | 8 | 11 | 19
  Unknown or Not Reported | 50 | 31 | 81
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 13 | 14 | 27
  Non-Hispanic | 92 | 88 | 180
  Unknown or Not Reported | 72 | 70 | 142

OUTCOME MEASURES:

1. Primary Outcome: SARS-CoV-2 Testing
Description: Yes/no indicator (coded 1 = yes, 0 = no) of whether or not person was tested for SARS-CoV-2 testing at syringe exchange visit, data collected from medical record
Time Frame: Immediate post intervention (i.e., same day)
Measure: Count of Participants; unit: Participants
Arm/Group | Connect2Test Intervention + Contingency Management | Contingency Management Alone
Number analyzed (Participants) | 177 | 172
Participants
  Was tested | 54 | 53
  Was not tested | 123 | 119
Statistical Analysis 1: Comparison: Connect2Test Intervention + Contingency Management vs Contingency Management Alone; Test type: Superiority; p = .944, Regression, Logistic — A priori threshold for statistical significance was p<.05; A multilevel logistic regression model was specified; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.62 to 1.56] — Contingency Management Alone coded as the reference group

2. Primary Outcome: SARS-CoV-2 Testing
Description: as for outcome 1
Time Frame: Up to 9-months after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Connect2Test Intervention + Contingency Management | Contingency Management Alone
Number analyzed (Participants) | 177 | 172
Participants
  Was tested | 46 | 46
  Was not tested | 131 | 126
Statistical Analysis 1: Comparison: Connect2Test Intervention + Contingency Management vs Contingency Management Alone; Test type: Superiority; p = .952, Regression, Logistic — A priori threshold for statistical significance was p<.05; A multilevel logistic regression model was specified; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.62 to 1.65] — Contingency Management Alone coded as the reference group

3. Secondary Outcome: COVID-19 Vaccination
Description: Yes/no indicator (coded 1 = yes, 0 = no) of whether or not person was vaccinated for COVID-19 at syringe exchange visit, data collected from vaccine records
Time Frame: Immediate post intervention (i.e., same day)
Measure: Count of Participants; unit: Participants
Arm/Group | Connect2Test Intervention + Contingency Management | Contingency Management Alone
Number analyzed (Participants) | 177 | 172
Participants
  Was vaccinated | 9 | 8
  Was not vaccinated | 168 | 164
Statistical Analysis 1: Comparison: Connect2Test Intervention + Contingency Management vs Contingency Management Alone; Test type: Superiority; p = .768, Regression, Logistic — A priori threshold for statistical significance was p<.05; A multilevel logistic regression model was specified; Odds Ratio (OR) = 1.16, 95% CI 2-sided [0.43 to 3.11] — Contingency Management Alone coded as the reference group

4. Secondary Outcome: COVID-19 Vaccination
Description: as for outcome 3
Time Frame: Up to 9-months after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Connect2Test Intervention + Contingency Management | Contingency Management Alone
Number analyzed (Participants) | 177 | 172
Participants
  Was vaccinated | 19 | 5
  Was not vaccinated | 158 | 167
Statistical Analysis 1: Comparison: Connect2Test Intervention + Contingency Management vs Contingency Management Alone; Test type: Superiority; p = .008, Regression, Logistic — A priori threshold for statistical significance was p<.05; A multilevel logistic regression model was specified; Odds Ratio (OR) = 3.96, 95% CI 2-sided [1.43 to 10.94] — Contingency Management Alone coded as the reference group

ADVERSE EVENTS:
Time Frame: Adverse event data was collected from completion of randomization through the 9-month follow-up period.
Arm/Group | Connect2Test Intervention + Contingency Management | Contingency Management Alone
All-Cause Mortality (participants affected / at risk) | 0/177 | 0/172
Serious Adverse Events (participants affected / at risk) | 0/177 | 0/172
Other Adverse Events (participants affected / at risk) | 0/177 | 0/172

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT05534061/Prot_002.pdf
  • Statistical Analysis Plan (2022-07-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT05534061/SAP_003.pdf
  • Informed Consent Form (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/61/NCT05534061/ICF_004.pdf